CLINICAL TRIAL: NCT02669368
Title: Effects of Magnesium Sulfate on Onset and Duration of Low Dose Rocuronium in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Magnesium Sulfate Effects on Onset and Duration of Low Dose Rocuronium in Patients Undergoing Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hamada Hamed, Dr., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01MgRo
Record Dates: First submitted 2016-01-25; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Muscle Relaxation
MeSH Terms: interventions — Magnesium Sulfate; Sodium Chloride; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Standard dose Rocuronium (Active Comparator): Pretreatment of saline 100ml then giving Rocuronium 0.6 mg/kg at induction of anesthesia.
  Interventions: Drug: Saline; Drug: Standard dose Rocuronium
- Low dose Rocuronium (Active Comparator): Pretreatment of saline 100ml then giving Rocuronium 0.45 mg/kg at induction of anesthesia.
  Interventions: Drug: Saline; Drug: Low dose Rocuronium
- Low dose Rocuronium + Magnesium Sulfate (Active Comparator): Pretreatment of Magnesium sulfate 30 mg/kg then giving Rocuronium 0.45 mg/kg at induction of anesthesia.
  Interventions: Drug: Magnesium Sulfate; Drug: Low dose Rocuronium

INTERVENTIONS:
Drug: Magnesium Sulfate — Patients in each group receive Magnesium sulfate 30 mg/kg in 0.9% normal saline (total volume 100 ml) intravenously for 5 min before induction of anesthesia
  Arms: Low dose Rocuronium + Magnesium Sulfate
Drug: Saline — Patients in each group receive 0.9% normal saline (total volume 100 ml) alone intravenously for 5 min before induction of anesthesia
  Arms: Low dose Rocuronium; Standard dose Rocuronium
Drug: Standard dose Rocuronium — 0.6 mg/kg of Rocuronium given with induction of anesthesia
  Arms: Standard dose Rocuronium
Drug: Low dose Rocuronium — 0.45 mg/kg of Rocuronium given with induction of anesthesia
  Arms: Low dose Rocuronium; Low dose Rocuronium + Magnesium Sulfate

SUMMARY:
This study aims to evaluate effects of magnesium sulfate on onset and duration of low dose rocuronium, intubation condition and surgical condition in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1 or 2.
* BMI of 25-34.9 kg/m2.
* Patients scheduled for laparoscopic cholecystectomy.

Exclusion Criteria:

* Severe respiratory or cardiac disease.
* Hepatic or renal function impairment.
* Neuromuscular disease.
* Patients on medications affecting neuromuscular function.
* Patients with known allergy to the drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The time of onset the action of Rocuronium | Time from injection of Rocuronium till T1 suppression more than 95% up to 10 minutes.
  by using the TOF watch nerve stimulator
The time at which Maximal suppression | Time from the injection of Rocuronium to T1 maximal suppression time (TOF=0) up to an hour.
  by using the TOF watch nerve stimulator
Reversal of Rocuronium | Time from injection of Rocuronium till reversal of T1 (TOF=25%) around an hour after induction of anesthesia
  by using the TOF watch nerve stimulator

SECONDARY OUTCOMES:
Intubation condition | Within 10 minutes after induction of anesthesia
  to score intubation condition on the basis of 6 items: Jaw relaxation, laryngoscopy, vocal cord position, moving of limbs, coughing & change in heart rate.
Surgical condition | During surgery
  to score a surgical condition according to 7 point likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Nawal Abdelaziz Gadelrab, Professor, Study Chair — Assiut University; Ola Mahmoud Wahba, Lecturer, Study Director — Assiut University Hospitals; Ahmed Hamada Hamed Amin, Resident, Principal Investigator — Assiut University Hospitals
Locations (1):
- Assiut University Hospitals, Asyut, Asyut Governorate, Egypt